CLINICAL TRIAL: NCT03289143
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy, and Safety Study of MTAU9937A in Patients With Prodromal to Mild Alzheimer's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Semorinemab in Patients With Prodromal to Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated during Open Label Extension period because analyses of placebo-controlled Blinded portion of study did not show any evidence of clinical efficacy or modulation of accumulation of tau PET signal at any of the doses studied.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GN39763; 2017-001800-31 (EudraCT Number)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer Disease; Brain Diseases; Dementia; Neurodegenerative Diseases; Neurocognitive Disorders
MeSH Terms: conditions — Alzheimer Disease; Brain Diseases; Dementia; Neurodegenerative Diseases; Neurocognitive Disorders | interventions — (18F)GTP1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Additional blinded personnel will include study site personnel who will evaluate participant status, contract research organization (CRO) personnel who will review case report forms (CRFs), and other sponsor agents (with the exception of the interactive voice or web-based response system [IxRS] vendor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 Semorinemab (Experimental)
  Interventions: Drug: Semorinemab; Drug: [18F]GTP1
- Dose 2 Semorinemab (Experimental)
  Interventions: Drug: Semorinemab; Drug: [18F]GTP1
- Dose 3 Semorinemab (Experimental)
  Interventions: Drug: Semorinemab; Drug: [18F]GTP1
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: [18F]GTP1

INTERVENTIONS:
Drug: Semorinemab — Participants will receive Semorinemab intravenously (IV).
  Other Names: RG6100; MTAU9937A; RO7105705
  Arms: Dose 1 Semorinemab; Dose 2 Semorinemab; Dose 3 Semorinemab
Drug: Placebo — Matching placebo doses of Semorinemab given intravenously (IV).
  Arms: Placebo
Drug: [18F]GTP1 — [18F]GTP1 will be administered as a solution for intravenous (IV) use, as part of positron emission tomography (PET) imaging.
  Other Names: RO6880276

SUMMARY:
This was a phase II, randomized, placebo-controlled, double-blind study to evaluate the efficacy and safety of Semorinemab in participants with prodromal to mild Alzheimer's disease. An optional 96-week open-label extension period was available to participants who completed the double-blind treatment period and who, in the judgment of the investigator, would potentially benefit from open-label Semorinemab treatment.

ELIGIBILITY:
Inclusion criteria

* Age between 50 and 80 years
* National Institute on Aging/Alzheimer's Association core clinical criteria for probable Alzheimer's disease (AD) dementia or mild cognitive impairment (prodromal AD)
* Evidence of the AD pathological process, by a positive amyloid assessment either on cerebrospinal fluid Aβ1-42 OR amyloid positron emission tomography (PET) scan. Historical amyloid PET scans may be accepted in some cases
* Mild AD symptomatology, as defined by a screening Mini-Mental State Examination score of >= 20 points and Clinical Dementia Rating (CDR) -Global Score of 0.5 or 1
* Abnormal memory function at screening
* Availability of a person with sufficient contact with the participant to be able to provide accurate information on the participant's cognitive and functional ability

Exclusion criteria

* Pregnant or breastfeeding
* Inability to tolerate magnetic resonance imaging (MRI) procedures or contraindication to MRI
* Contraindications to both PET imaging and lumbar dural puncture (must be able to undergo at least one of these procedures to be eligible)
* Residence in a skilled nursing facility
* Any serious medical condition or abnormality in clinical laboratory tests that remains abnormal on retest and, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or bias the assessment of the clinical or mental status of the participant to a significant degree
* Any evidence of a condition other than AD that may affect cognition
* Alcohol or substance abuse within the past 2 years
* Use of any experimental therapy within 90 days or 5 half-lives prior to screening, whichever is greater and any passive immunotherapy (immunoglobulin) against tau, except use of RO7105705 in Genentech Study GN39058, as long as the last dose was at least 90 days prior to screening
* Use of any passive immunotherapy (immunoglobulin) against Aβ, unless the last dose was at least 1 year prior to screening and any active immunotherapy (vaccine) that is under evaluation to prevent or postpone cognitive decline
* Any previous treatment with medications specifically intended to treat Parkinsonian symptoms or any other neurodegenerative disorder within 1 year of screening
* Systemic immunosuppressive therapy within 12 months of screening through the entire study period
* Typical antipsychotic or neuroleptic medication within 6 months of screening
* Daily treatment with any of the following classes of medication, except for intermittent short-term use, which is permitted except within 2 days or 5 half-lives (whichever is longer) prior to any COA: atypical antipsychotics, opiates or opioids, benzodiazepines, barbiturates, hypnotics, or any medication with clinically significant centrally-acting antihistamine or anticholinergic activity
* Stimulant medications, unless the dose has been stable within the 6 months prior to screening and is expected to be stable throughout the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (133):
- United States (43):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Clinical Trials, Glendale, California
  - University of California Irvine, Irvine, California
  - Pharmacology Research Inst, Newport Beach, California
  - Stanford Neuroscience Health Center (SNHC), Palo Alto, California
  - Pacific Research Network - PRN, San Diego, California
  - Neurological Research Inst, Santa Monica, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - Invicro, a Konica Minolta company, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - KI Health Partners, LLC; New England Institute for Clinical Research, Stamford, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - JEM Research LLC, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Compass Research East, LLC, Orlando, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University; Global Health, Atlanta, Georgia
  - Rush Alzheimer's Disease Cntr., Chicago, Illinois
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Eastern Maine Medical Center, Bangor, Maine
  - Brigham & Women's Hosp; TIMI Study Grp, Boston, Massachusetts
  - Alzheimers Disease Center, Quincy, Massachusetts
  - Health Partners Institute for Education and Research, Saint Paul, Minnesota
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Albany Medical College; Neurology, Albany, New York
  - Empire Neurology PC; MS Center of Northeastern NY, Latham, New York
  - Columbia Univ Medical Center, New York, New York
  - University of Rochester; AD-CARE, Rochester, New York
  - Summit Research Network Inc., Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Neurology Clinic PC, Cordova, Tennessee
  - New Orleans Center For Clinical Research, Knoxville, Tennessee
  - Clinical Neuroscience Research Associates, Inc., Bennington, Vermont
- Australia (8):
  - St Vincents Medical Centre, Darlinghurst, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - Queensland University of Technology, Mermaid Waters, Queensland
  - Eastern Clinical Research Unit; Pharmacy, Box Hill, Victoria
  - HammondCare Aged Psychiatry Clinical Trials, Malvern, Victoria
  - The Alfred Hospital, Melbourne; Thrombosis and Haemostasis Unit, Melbourne, Victoria
  - Neuro Trials Victoria, Noble Park, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (4):
  - UZ Brussel, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Delta Campus Westlaan, Roeselare
- Canada (8):
  - JBN Medical Diagnostic Services; Clinical Trials Division, Burlington, Ontario
  - Parkwood Institute, Mental Health Care Building, London, Ontario
  - Elisabeth Bruyere Hospital, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Centre for Memory and Aging, Toronto, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Recherches Neuro-Hippocame, Gatineau, Quebec
- Denmark (2):
  - Center For Clinical and Basic Research (Ccbr); Site Management Organisation, Aalborg
  - CCBR - Vejle - DK, Vejle
- France (12):
  - Groupe Hospitalier Pellegrin; Service de Neurologie - 3ème étage, Bordeaux
  - Hopital Neurologique Pierre Wertheimer, Bron
  - Hopital Roger Salengro, Lille
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - Hopital Fernand Widal Centre, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - CHU Rennes, Rennes
  - CHU Hautepierre; ACTR Association Recherche Clinique Rhumatologie, Strasbourg
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg
  - Hopital de La Grave, Toulouse
  - Hopital des Charpennes, Villeurbanne
- Germany (11):
  - Klinikum Bayreuth; Krankenhaus Hohe Warte, Bayreuth
  - Praxis Dr. med. Volker Shumann, Berlin
  - Studienambulanz emovis GmbH; St. Joseph Krankenhaus, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Neurologisch-psychiatrische Praxis am Brosepark, Berlin
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Klinikum rechts der Isar der TU München; Klinik & Poliklinik für Neurologie, München
  - ZNS Siegen im MVZ Weidenau, Siegen
  - Universitätsklinik Tübingen; Psychiatrie und Psychotherapie, Tübingen
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
- Italy (7):
  - Az. Osp. C. Panico; Rep. Ematologia E Trapianto, Tricase - LE, Apulia
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratell;Neurologia, Rome, Lazio
  - Azienda Ospedaliero Universitaria San Martino; Dip. di Neuroscienze Oftalmologia e Genetica, Genoa, Liguria
  - IRCCS Centro San Giovanni di Dio FBF, Brescia, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - IRCCS Neuromed; Neurologia I-Centro studio e cura delle demenze e UVA, Pozzilli, Molise
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Brain Research Center B.V, Amsterdam
- Poland (12):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - PALLMED Sp. z o.o. prowadząca NZOZ DOM SUE RYDER, Bydgoszcz
  - M.A. - LEK A.M.Maciejowscy SC., Katowice
  - Novo-Med Zielinski i wspolnicy Sp. j., Katowice
  - Malopolskie Centrum Medyczne, Krakow
  - NEURO - KARD Ośrodek Badań Klinicznych, Poznan
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - EroMedis, Szczecin
  - AMED Medical Center, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - NZOZ WCA, Wroclaw
- Spain (15):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Clinica Universitaria de Navarra; Servicio de Neurología, Pamplona, Navarre
  - Hospital Virgen del Puerto, Plasencia, Palencia
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Hospital Perpetuo Socorro, Servicio de Geriatria, Albacete
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundación ACE; Servicio de Neurología, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Neurologia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital de Cantoblanco; Servicio de Geriatria, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Dr. Peset; Servicio de Neurologia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (5):
  - Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset Kalmar; Oncology, Kalmar
  - Skane University Hospital Malmo/Lund, Dept.of Hematology and Coagulation Disorders, Malmo
  - Sahlgrenska Univ Hospital Mölndal; Department of Nephrology, Mölndal
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- United Kingdom (4):
  - Glasgow Memory Clinic, Glasgow
  - RE:Cognition Health, London
  - The National Hospital for Neurology & Neurosurgery, London
  - Re:Cognition Health Guildford, Surrey

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Schauer SP, Toth B, Lee J, Honigberg LA, Ramakrishnan V, Jiang J, Kollmorgen G, Bayfield A, Wild N, Hoffman J, Ceniceros R, Dolton M, Bohorquez SMS, Hoogenraad CC, Wildsmith KR, Teng E, Monteiro C, Anania V, Yeh FL. Pharmacodynamic effects of semorinemab on plasma and CSF biomarkers of Alzheimer's disease pathophysiology. Alzheimers Dement. 2024 Dec;20(12):8855-8866. doi: 10.1002/alz.14346. Epub 2024 Nov 8. PMID 39513754
- [Derived] Sanabria Bohorquez SM, Baker S, Manser PT, Tonietto M, Galli C, Wildsmith KR, Zou Y, Kerchner GA, Weimer R, Teng E. Evaluation of partial volume correction and analysis of longitudinal [18F]GTP1 tau PET imaging in Alzheimer's disease using linear mixed-effects models. Front Neuroimaging. 2024 Mar 28;3:1355402. doi: 10.3389/fnimg.2024.1355402. eCollection 2024. PMID 38606196
- [Derived] Teng E, Li Y, Manser PT, Pickthorn K, Butcher BD, Blendstrup M, Randolph C, Sikkes SAM. Cross-sectional and longitudinal assessments of function in prodromal-to-mild Alzheimer's disease: A comparison of the ADCS-ADL and A-IADL-Q scales. Alzheimers Dement (Amst). 2023 Jun 13;15(2):e12452. doi: 10.1002/dad2.12452. eCollection 2023 Apr-Jun. PMID 37325545
- [Derived] Teng E, Manser PT, Shah M, Pickthorn K, Hu N, Djakovic S, Swendsen H, Blendstrup M, Faccin G, Ostrowitzki S, Sink KM. The Use of Episodic Memory Tests for Screening in Clinical Trials for Early Alzheimer's Disease: A Comparison of the Free and Cued Selective Reminding Test (FCSRT) and the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). J Prev Alzheimers Dis. 2023;10(1):41-49. doi: 10.14283/jpad.2022.101. PMID 36641609
- [Derived] Teng E, Manser PT, Pickthorn K, Brunstein F, Blendstrup M, Sanabria Bohorquez S, Wildsmith KR, Toth B, Dolton M, Ramakrishnan V, Bobbala A, Sikkes SAM, Ward M, Fuji RN, Kerchner GA; Tauriel Investigators. Safety and Efficacy of Semorinemab in Individuals With Prodromal to Mild Alzheimer Disease: A Randomized Clinical Trial. JAMA Neurol. 2022 Aug 1;79(8):758-767. doi: 10.1001/jamaneurol.2022.1375. PMID 35696185

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a double-blind treatment period and an optional open-label extension (OLE) period. OLE period was available to participants who completed the double-blind treatment period and who, in the judgment of the investigator, would potentially benefit from open-label semorinemab treatment.
Groups:
- Placebo Double Blind Period: Matching placebo dose of Semorinemab was administered intravenously in the double-blind treatment period.
- Dose 1 Semorinemab Double Blind Period: Semorinemab was administered intravenously at dose 1 in the double-blind treatment period.
- Dose 2 Semorinemab Double Blind Period: Semorinemab was administered intravenously at dose 2 in the double-blind treatment period.
- Dose 3 Semorinemab Double Blind Period: Semorinemab was administered intravenously at dose 3 in the double-blind treatment period.
Period: Overall Study
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Started | 135 | 94 | 136 | 92
Completed | 1 | 0 | 2 | 0
Not Completed | 134 | 94 | 134 | 92
Not completed — Caregiver Unavailability | 1 | 1 | 0 | 0
Not completed — Research Department Closure | 0 | 0 | 1 | 0
Not completed — Caregiver and Participant Withdrew Consent | 0 | 0 | 1 | 0
Not completed — Medical Monitor Decision | 1 | 0 | 0 | 0
Not completed — Participant Non-Compliance | 0 | 0 | 1 | 0
Not completed — Drug Interrupted for Too Long Due to Prohibited Med | 0 | 0 | 1 | 0
Not completed — Participant Non Compliance With Concomitant Medications | 0 | 0 | 1 | 0
Not completed — Caregiver Passed Away | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 2 | 2
Not completed — Protocol Deviation | 2 | 1 | 3 | 1
Not completed — Study Terminated By Sponsor | 101 | 75 | 100 | 69
Not completed — Withdrawal by Subject | 14 | 6 | 14 | 12
Not completed — Adverse Event | 10 | 7 | 6 | 5
Not completed — Death | 2 | 0 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0
Not completed — Participant No Longer Has Study Partner | 0 | 0 | 0 | 1
Not completed — Withdrawal by Caregiver | 0 | 1 | 0 | 0
Not completed — Caregiver Passed Away & Family Moved Out of State | 0 | 0 | 1 | 0
Not completed — Absence of Consistent and Reliable Caregiver | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period | Total
Number analyzed (Participants) | 135 | 94 | 136 | 92 | 457
Age, Continuous [Mean (Standard Deviation); unit: Year] | 69.7 (7.3) | 70.2 (6.7) | 69.3 (7.1) | 69.6 (6.7) | 69.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 51 | 79 | 48 | 253
  Male | 60 | 43 | 57 | 44 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5 | 3 | 13
  Not Hispanic or Latino | 126 | 80 | 125 | 79 | 410
  Unknown or Not Reported | 8 | 10 | 6 | 10 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 1 | 1 | 4
  White | 129 | 83 | 128 | 82 | 422
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 4 | 6 | 5 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the CDR-SB
Description: The Clinical Dementia Rating-Sum of Boxes (CDR-SB) rates impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment = 0, questionable impairment = 0.5 and mild, moderate and severe impairment = 1, 2 and 3 respectively. The score range is from 0 to 18 with a high score indicating a high disease severity. The difference in mean change from Baseline to Week 73 between Semorinemab doses and Placebo treated participants was estimated. The difference in mean change from Baseline to Week 73 between Semorinemab doses and Placebo treated participants was estimated.
Time Frame: Baseline and 73 Weeks
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of study drug and had at least one postbaseline primary efficacy Clinical Dementia Rating-Sum of Boxes (CDR-SB) measurement.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Number analyzed (Participants) | 105 | 77 | 113 | 74
Units on a scale | 2.19 (0.226) | 2.36 (0.268) | 2.36 (0.222) | 2.41 (0.27)
Statistical Analysis 1: Comparison: Placebo Double Blind Period vs Dose 1 Semorinemab Double Blind Period; Test type: Superiority; p = 0.6147, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 2: Comparison: Placebo Double Blind Period vs Dose 2 Semorinemab Double Blind Period; Test type: Superiority; p = 0.5778, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 3: Comparison: Placebo Double Blind Period vs Dose 3 Semorinemab Double Blind Period; Test type: Superiority; p = 0.5136, Mixed-effect Model Repeated Measures — Unadjusted

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with at least one adverse event
Time Frame: Up to the data cutoff date 15 January 2021 (up to approximately 39 months)
Population: The safety-evaluable population included all participants who were randomly allocated and received at least one dose of study drug (MTAU9937A or placebo) during the double-blind treatment period with treatment groups defined according to actual treatment received.
Measure: Number; unit: Percentage of participants
Groups:
- Dose 2 Semorinemab Open Label Extension Period: Semorinemab was administered intravenously at dose 2 in the open-label extension period.
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period | Dose 2 Semorinemab Open Label Extension Period
Number analyzed (Participants) | 130 | 89 | 132 | 90 | 360
Percentage of participants | 93.1 | 88.8 | 94.7 | 92.2 | 47.5

3. Secondary Outcome: Change From Baseline on the Repeatable Battery for Assessment of Neuropsychological Status (RBANS)
Description: The RBANS is a validated neuropsychological assessment has been shown to be a useful tool in both clinical and research settings. The RBANS consists of ten subtests that are combined to provide five indices, one for each of the five domains tested (immediate memory, visuospatial/constructional, language, attention, and delayed memory). Scores range from 40 to 160 and a higher score indicates better cognitive functioning. A decrease in the outcome measure from baseline corresponds to disease worsening. The difference in mean change from Baseline to Week 73 between Semorinemab doses and Placebo treated participants was estimated.
Time Frame: Baseline and 73 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Number analyzed (Participants) | 87 | 62 | 93 | 63
Score on a scale | -5.53 (0.787) | -5.25 (0.93) | -4.62 (0.765) | -6.15 (0.926)
Statistical Analysis 1: Comparison: Placebo Double Blind Period vs Dose 1 Semorinemab Double Blind Period; Test type: Superiority; p = 0.8198, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 2: Comparison: Placebo Double Blind Period vs Dose 2 Semorinemab Double Blind Period; Test type: Superiority; p = 0.3961, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 3: Comparison: Placebo Double Blind Period vs Dose 3 Semorinemab Double Blind Period; Test type: Superiority; p = 0.6043, Mixed-effect Model Repeated Measures — Unadjusted

4. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Assessment Scale-Cognitive Subscale 13 (ADAS-Cog-13) Subscale Score
Description: The ADAS-Cog-13 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Most of these are assessed by tests although some are rated by the clinician on a 5-point scale. The ADAS-Cog-13 is the ADAS-Cog-11 with 2 further items: delayed word recall and total digit cancellation. The score range for ADAS-Cog-13 is from 0 to 85 with high scores representing severe dysfunction. The difference in mean change from Baseline to Week 73 between Semorinemab doses and Placebo treated participants was estimated.
Time Frame: Baseline and 73 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Number analyzed (Participants) | 94 | 67 | 97 | 66
Score on a scale | 6.56 (0.777) | 8.68 (0.937) | 6 (0.769) | 7.58 (0.932)
Statistical Analysis 1: Comparison: Placebo Double Blind Period vs Dose 1 Semorinemab Double Blind Period; Test type: Superiority; p = 0.0783, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 2: Comparison: Placebo Double Blind Period vs Dose 2 Semorinemab Double Blind Period; Test type: Superiority; p = 0.6010, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 3: Comparison: Placebo Double Blind Period vs Dose 3 Semorinemab Double Blind Period; Test type: Superiority; p = 0.3961, Mixed-effect Model Repeated Measures — Unadjusted

5. Secondary Outcome: Change From Baseline on the Amsterdam Instrumental Activity of Daily Living (iADL) Questionnaire
Description: The Amsterdam iADL questionnaire is an informant-based instrument for measuring iADL problems in participants with dementia. This instrument consists of 70 items, scored on a 5-point scale, that uses item response theory for scoring. Items presented to the informant are tailored to responses to earlier items; thus each administration of the Amsterdam iADL may consist of less than the total of 70 items. The resulting score ranges from 20 to 80 with lower scores indicating poorer performance. A decrease in the outcome measure from baseline corresponds to disease worsening. The difference in mean change from Baseline to Week 73 between Semorinemab doses and Placebo treated participants was estimated.
Time Frame: Baseline and 73 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Number analyzed (Participants) | 95 | 70 | 109 | 67
Score on a scale | -6.59 (0.856) | -6.55 (0.999) | -6.92 (0.824) | -7.31 (1.013)
Statistical Analysis 1: Comparison: Placebo Double Blind Period vs Dose 1 Semorinemab Double Blind Period; Test type: Superiority; p = 0.9749, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 2: Comparison: Placebo Double Blind Period vs Dose 2 Semorinemab Double Blind Period; Test type: Superiority; p = 0.7718, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 3: Comparison: Placebo Double Blind Period vs Dose 3 Semorinemab Double Blind Period; Test type: Superiority; p = 0.5789, Mixed-effect Model Repeated Measures — Unadjusted

6. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Cooperative Study Group-Activities of Daily Living Inventory
Description: The ADCS-ADL (Alzheimer's Disease Cooperative Study-Activities of Daily Living) is the scale most widely used to assess functional outcomes in participants with AD. The ADCS-ADL covers both basic ADL (e.g., eating and toileting) and more complex 'instrumental' ADL or iADL (e.g., using the telephone, managing finances and preparing a meal). The ADCS-ADL consists of 23 questions with a score range of 0 to 78 where a higher score represents better function. The difference in mean change from Baseline to Week 73 between Semorinemab doses and Placebo treated participants was estimated.
Time Frame: Baseline and 73 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Number analyzed (Participants) | 104 | 76 | 112 | 74
Score on a scale | -8.55 (0.996) | -9.52 (1.179) | -7.75 (0.986) | -7.99 (1.183)
Statistical Analysis 1: Comparison: Placebo Double Blind Period vs Dose 1 Semorinemab Double Blind Period; Test type: Superiority; p = 0.5235, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 2: Comparison: Placebo Double Blind Period vs Dose 2 Semorinemab Double Blind Period; Test type: Superiority; p = 0.5612, Mixed-effect Model Repeated Measures — Unadjusted
Statistical Analysis 3: Comparison: Placebo Double Blind Period vs Dose 3 Semorinemab Double Blind Period; Test type: Superiority; p = 0.7130, Mixed-effect Model Repeated Measures — Unadjusted

7. Secondary Outcome: Serum Concentrations of Semorinemab at Specified Timepoints
Description: Serum concentrations of Semorinemab at specified timepoints.
Time Frame: Up to 109 weeks
Population: The PK-evaluable population is defined as patients who received Semorinemab treatment and had at least one measureable PK concentration.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Dose 1 Semorinemab Double Blind and Open Label Extension Periods: Semorinemab was administered intravenously at dose 1 in the double-blind treatment period. Optional Open Label Extension was available to participants who completed the double-blind treatment period and who, in the judgment of the investigator, would potentially benefit from open-label extension.
- Dose 2 Semorinemab Double Blind and Open Label Extension Periods: Semorinemab was administered intravenously at dose 2 in the double-blind treatment period. Optional Open Label Extension was available to participants who completed the double-blind treatment period and who, in the judgment of the investigator, would potentially benefit from open-label extension.
- Dose 3 Semorinemab Double Blind and Open Label Extension Periods: Semorinemab was administered intravenously at dose 3 in the double-blind treatment period. Optional Open Label Extension was available to participants who completed the double-blind treatment period and who, in the judgment of the investigator, would potentially benefit from open-label extension.
Arm/Group | Dose 1 Semorinemab Double Blind and Open Label Extension Periods | Dose 2 Semorinemab Double Blind and Open Label Extension Periods | Dose 3 Semorinemab Double Blind and Open Label Extension Periods
Number analyzed (Participants) | 89 | 132 | 90
ug/mL
  Week 1, 0-4 Hours Predose: number analyzed (Participants) | 87 | 132 | 90
  Week 1, 0-4 Hours Predose | NA (NA) — Not reportable. Below the level of detection. | NA (NA) — Not reportable. Below the level of detection. | NA (NA) — Not reportable. Below the level of detection.
  Week 1, 1 Hour Postdose: number analyzed (Participants) | 87 | 132 | 90
  Week 1, 1 Hour Postdose | 472 (131) | 1580 (496) | 2690 (689)
  Week 1, 2 Hours Postdose: number analyzed (Participants) | 86 | 130 | 90
  Week 1, 2 Hours Postdose | 476 (123) | 1510 (419) | 2600 (707)
  Week 1, 4 Hours postdose: number analyzed (Participants) | 86 | 128 | 89
  Week 1, 4 Hours postdose | 463 (135) | 1370 (405) | 2570 (785)
  Week 3, 0-4 hours Predose: number analyzed (Participants) | 89 | 131 | 89
  Week 3, 0-4 hours Predose | 184 (52.7) | 601 (211) | 1100 (449)
  Week 3, 30 min Post dose: number analyzed (Participants) | 88 | 130 | 88
  Week 3, 30 min Post dose | 718 (198) | 2320 (581) | 4190 (1010)
  Week 5, 0-4 Hours Predose: number analyzed (Participants) | 88 | 131 | 87
  Week 5, 0-4 Hours Predose | 318 (81.5) | 955 (256) | 1920 (614)
  Week 5, 30 min Postdose: number analyzed (Participants) | 86 | 130 | 85
  Week 5, 30 min Postdose | 908 (508) | 2780 (695) | 4860 (1250)
  Week 9, 0-4 hours Predose: number analyzed (Participants) | 88 | 130 | 83
  Week 9, 0-4 hours Predose | 344 (128) | 961 (288) | 1840 (513)
  Week 9, 30 Minutes Postdose: number analyzed (Participants) | 89 | 129 | 85
  Week 9, 30 Minutes Postdose | 889 (321) | 2790 (757) | 4960 (1270)
  Week 13, 0-4 Hours Predose: number analyzed (Participants) | 87 | 128 | 86
  Week 13, 0-4 Hours Predose | 360 (105) | 1060 (333) | 1910 (545)
  Week 13, 30 Minutes Postdose: number analyzed (Participants) | 86 | 127 | 86
  Week 13, 30 Minutes Postdose | 998 (896) | 2900 (668) | 4880 (1250)
  Week 17: number analyzed (Participants) | 0 | 0 | 1
  Week 17 |  |  | 1750 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Week 17, 0-4 Hours Predose: number analyzed (Participants) | 84 | 127 | 83
  Week 17, 0-4 Hours Predose | 386 (116) | 1040 (316) | 1890 (522)
  Week 17, 30 Minutes Postdose: number analyzed (Participants) | 84 | 126 | 86
  Week 17, 30 Minutes Postdose | 819 (242) | 2930 (902) | 4770 (1270)
  Week 33, 0-4 Hours Predose: number analyzed (Participants) | 83 | 126 | 83
  Week 33, 0-4 Hours Predose | 404 (134) | 960 (277) | 2050 (648)
  Week 33, 30 Minutes Postdose: number analyzed (Participants) | 82 | 126 | 80
  Week 33, 30 Minutes Postdose | 801 (260) | 2540 (853) | 4800 (1200)
  Week 49, 0-4 Hours Predose: number analyzed (Participants) | 78 | 119 | 79
  Week 49, 0-4 Hours Predose | 377 (105) | 1060 (332) | 2160 (605)
  Week 49, 30 Minutes Postdose: number analyzed (Participants) | 77 | 117 | 80
  Week 49, 30 Minutes Postdose | 871 (260) | 2810 (967) | 4960 (1030)
  Week 65: number analyzed (Participants) | 0 | 0 | 1
  Week 65 |  |  | 2100 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category.
  Week 65, 0-4 Hours Predose: number analyzed (Participants) | 67 | 101 | 66
  Week 65, 0-4 Hours Predose | 405 (127) | 1170 (276) | 2020 (681)
  Week 65, 30 Minutes Postdose: number analyzed (Participants) | 67 | 100 | 67
  Week 65, 30 Minutes Postdose | 963 (401) | 2930 (830) | 4710 (1450)
  Week 73: number analyzed (Participants) | 71 | 104 | 69
  Week 73 | 327 (154) | 1030 (451) | 1830 (752)
  Week 73, 0-4 Hours Predose: number analyzed (Participants) | 0 | 1 | 0
  Week 73, 0-4 Hours Predose |  | 382 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. |
  Week 73, 1 Hour Postdose: number analyzed (Participants) | 0 | 1 | 0
  Week 73, 1 Hour Postdose |  | 1910 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. |
  Week 73, 2 Hours Postdose: number analyzed (Participants) | 0 | 1 | 0
  Week 73, 2 Hours Postdose |  | 1740 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. |
  Week 73, 4 Hours Postdose: number analyzed (Participants) | 0 | 1 | 0
  Week 73, 4 Hours Postdose |  | 1710 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. |
  Week 77 OLE, 0-4 Hours Predose: number analyzed (Participants) | 13 | 20 | 13
  Week 77 OLE, 0-4 Hours Predose | 180 (71.0) | 724 (167) | 1030 (345)
  Week 77 OLE, 1 hour Postdose: number analyzed (Participants) | 12 | 20 | 12
  Week 77 OLE, 1 hour Postdose | 1700 (523) | 2460 (868) | 2670 (707)
  Week 77 OLE, 2 hours Postdose: number analyzed (Participants) | 13 | 20 | 13
  Week 77 OLE, 2 hours Postdose | 1830 (552) | 2270 (442) | 2510 (579)
  Week 77 OLE, 4 hours Postdose: number analyzed (Participants) | 11 | 20 | 12
  Week 77 OLE, 4 hours Postdose | 1850 (516) | 2270 (480) | 2790 (558)
  Week 93 OLE, 0-4 Hours Pre-dose: number analyzed (Participants) | 2 | 2 | 4
  Week 93 OLE, 0-4 Hours Pre-dose | 632 (37.5) | 1040 (113) | 1290 (307)
  Week 93 OLE, 30 Minutes Postdose: number analyzed (Participants) | 2 | 2 | 4
  Week 93 OLE, 30 Minutes Postdose | 1920 (431) | 2570 (91.9) | 2880 (492)
  Week 109 OLE, 0-4 Hours Predose: number analyzed (Participants) | 0 | 1 | 0
  Week 109 OLE, 0-4 Hours Predose |  | 1270 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. |
  Week 109 OLE, 30 Minutes Postdose: number analyzed (Participants) | 0 | 1 | 0
  Week 109 OLE, 30 Minutes Postdose |  | 3330 (NA) — Data not reported because SD was non-estimable since only 1 participant was evaluated for this category. |

8. Secondary Outcome: Presence of Anti-drug Antibodies During the Study Relative to Their Presence at Baseline
Description: Presence of anti-drug antibodies during the study relative to their presence at baseline.
Time Frame: Up to 109 weeks
Population: The immunogenicity analyses will include participants with at least one predose and one postdose ADA assessment, with participants grouped according to treatment arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period
Number analyzed (Participants) | 130 | 89 | 132 | 90
Percentage of participants
  Baseline: number analyzed (Participants) | 127 | 87 | 132 | 90
  Baseline | 0 | 0 | 0 | 0
  Post-baseline: number analyzed (Participants) | 0 | 86 | 128 | 88
  Post-baseline |  | 0 | 0 | 0

9. Primary Outcome: Change From Baseline on the C-SSRS
Description: Categories are as defined in the Classification Algorithm for Suicide Assessment (CASA) based on the Columbia Suicide Severity Rating Scale (C-SSRS) questionnaire. SI1: Passive category is "Wish to be dead", SI2: Active-Nonspecific (no method, intent or plan), SI3: Active-Method, but no intent or Plan, SI4: Active-Method and intent, but no plan in C-SSRS. The worst post-baseline suicidal ideation is the highest across post-baseline visits, with highest as SI5 and lowest as SI1. Percentages are based on the total number of subjects in a treatment group. Baseline is the last observation prior to initiation of study drug.
Time Frame: Baseline to data cutoff date 15 January 2021 (up to approximately 39 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period | Dose 2 Semorinemab Open Label Extension Period
Number analyzed (Participants) | 130 | 89 | 132 | 90 | 360
Participants
  Missing/No Events | 1 | 1 | 2 | 0 | 3
  Missing/SI1 | 0 | 0 | 0 | 0 | 0
  Missing/SI2 | 0 | 0 | 0 | 0 | 0
  Missing/SI3 | 0 | 0 | 0 | 0 | 0
  Missing/SI4 | 0 | 0 | 0 | 0 | 0
  Missing/Missing | 0 | 0 | 0 | 0 | 0
  No Event/No Event | 119 | 80 | 123 | 83 | 336
  No Event/SI1 | 3 | 3 | 2 | 4 | 5
  No Event/ SI2 | 0 | 1 | 1 | 0 | 1
  No Event/SI3 | 0 | 0 | 0 | 0 | 0
  No Event/ SI4 | 0 | 0 | 0 | 0 | 0
  No Event/ Missing | 1 | 0 | 0 | 1 | 1
  SI1/No Event | 3 | 3 | 1 | 1 | 8
  SI1/SI1 | 0 | 0 | 0 | 0 | 1
  SI1/SI2 | 1 | 0 | 0 | 0 | 0
  SI1/SI3 | 0 | 0 | 0 | 0 | 0
  SI1/SI4 | 1 | 0 | 0 | 0 | 0
  SI1/Missing | 0 | 0 | 0 | 0 | 0
  SI2/No Event | 0 | 1 | 2 | 0 | 1
  SI2/SI1 | 0 | 0 | 1 | 0 | 2
  SI2/SI2 | 0 | 0 | 0 | 1 | 0
  SI2/SI3 | 0 | 0 | 0 | 0 | 0
  SI2/SI4 | 0 | 0 | 0 | 0 | 0
  SI2/Missing | 0 | 0 | 0 | 0 | 0
  SI3/No Event | 1 | 0 | 0 | 0 | 1
  SI3/SI1 | 0 | 0 | 0 | 0 | 0
  SI3/SI2 | 0 | 0 | 0 | 0 | 0
  SI3/SI3 | 0 | 0 | 0 | 0 | 0
  SI3/SI4 | 0 | 0 | 0 | 0 | 0
  SI3/Missing | 0 | 0 | 0 | 0 | 0
  SI4/No Event | 0 | 0 | 0 | 0 | 0
  SI4/SI1 | 0 | 0 | 0 | 0 | 0
  SI4/SI2 | 0 | 0 | 0 | 0 | 0
  SI4/SI3 | 0 | 0 | 0 | 0 | 1
  SI4/Missing | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Other Abnormal MRI Findings
Description: Other abnormal MRI findings by visit. For the Double Blind Period, baseline is defined as last results prior to initiation of study drug. For the Open Label Extension Period, baseline is defined as last results prior to entering the open label period.
Time Frame: Baseline, Week 9, Week 49, Week 73, Study Treatment Discontinuation, and Week 89
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period | Dose 2 Semorinemab Open Label Extension Period
Number analyzed (Participants) | 135 | 94 | 136 | 92 | 360
Number of participants
  Cerebrovascular Pathology, Baseline | 3 | 0 | 2 | 1 | 5
  CNS Trauma, Baseline | 0 | 0 | 0 | 1 | 1
  Intracranial Tumor, Baseline | 0 | 0 | 3 | 2 | 4
  Lacunar Infarct, Baseline | 13 | 3 | 11 | 6 | 23
  Superficial Hemosiderosis, Baseline | 3 | 0 | 2 | 0 | 7
  Territorial Infarct, Baseline | 3 | 1 | 0 | 0 | 4
  Vasogenic Edema/Sulcal Effusion, Baseline | 0 | 0 | 0 | 0 | 0
  Cerebrovascular Pathology, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Cerebrovascular Pathology, Week 9 | 0 | 1 | 0 | 0 |
  CNS Trauma, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  CNS Trauma, Week 9 | 0 | 0 | 0 | 0 |
  Intracranial Tumor, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Intracranial Tumor, Week 9 | 0 | 0 | 0 | 0 |
  Lacunar Infarct, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Lacunar Infarct, Week 9 | 0 | 1 | 0 | 0 |
  Superficial Hemosiderosis, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Superficial Hemosiderosis, Week 9 | 3 | 0 | 0 | 1 |
  Territorial Infarct, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Territorial Infarct, Week 9 | 0 | 0 | 0 | 0 |
  Vasogenic Edema/Sulcal Effusion, Week 9: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Vasogenic Edema/Sulcal Effusion, Week 9 | 0 | 0 | 1 | 0 |
  Cerebrovascular Pathology, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Cerebrovascular Pathology, Week 49 | 0 | 0 | 0 | 0 |
  CNS Trauma, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  CNS Trauma, Week 49 | 0 | 0 | 0 | 0 |
  Intracranial Tumor, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Intracranial Tumor, Week 49 | 0 | 0 | 0 | 0 |
  Lacunar Infarct, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Lacunar Infarct, Week 49 | 0 | 0 | 0 | 0 |
  Superficial Hemosiderosis, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Superficial Hemosiderosis, Week 49 | 1 | 1 | 1 | 0 |
  Territorial Infarct, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Territorial Infarct, Week 49 | 0 | 0 | 0 | 0 |
  Vasogenic Edema/Sulcal Effusion, Week 49: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Vasogenic Edema/Sulcal Effusion, Week 49 | 0 | 0 | 0 | 0 |
  Cerebrovascular Pathology, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Cerebrovascular Pathology, Week 73 | 0 | 0 | 0 | 0 |
  CNS Trauma, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  CNS Trauma, Week 73 | 0 | 0 | 0 | 0 |
  Intracranial Tumor, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Intracranial Tumor, Week 73 | 1 | 0 | 0 | 0 |
  Lacunar Infarct, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Lacunar Infarct, Week 73 | 0 | 1 | 0 | 0 |
  Superficial Hemosiderosis, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Superficial Hemosiderosis, Week 73 | 0 | 1 | 0 | 1 |
  Territorial Infarct, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Territorial Infarct, Week 73 | 0 | 0 | 0 | 0 |
  Vasogenic Edema/Sulcal Effusion, Week 73: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Vasogenic Edema/Sulcal Effusion, Week 73 | 1 | 0 | 0 | 0 |
  Cerebrovascular Pathology, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Cerebrovascular Pathology, Study Treatment Early Discontinuation | 0 | 0 | 0 | 0 |
  CSN Trauma, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  CSN Trauma, Study Treatment Early Discontinuation | 0 | 0 | 0 | 0 |
  Intracranial Tumor, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Intracranial Tumor, Study Treatment Early Discontinuation | 0 | 0 | 0 | 0 |
  Lucunar Infarct, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Lucunar Infarct, Study Treatment Early Discontinuation | 1 | 0 | 0 | 0 |
  Superficial Hemosiderosis, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Superficial Hemosiderosis, Study Treatment Early Discontinuation | 1 | 0 | 0 | 0 |
  Territorial Infarct, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Territorial Infarct, Study Treatment Early Discontinuation | 0 | 0 | 0 | 0 |
  Vasogenic Edema/Sulcal Effusion, Study Treatment Early Discontinuation: number analyzed (Participants) | 135 | 94 | 136 | 92 | 0
  Vasogenic Edema/Sulcal Effusion, Study Treatment Early Discontinuation | 0 | 0 | 0 | 0 |
  Cerebrovascular Pathology, Week 89 Open Label Extension (OLE): number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  Cerebrovascular Pathology, Week 89 Open Label Extension (OLE) |  |  |  |  | 0
  CNS Trauma, Week 89 OLE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  CNS Trauma, Week 89 OLE |  |  |  |  | 0
  Intracranial Tumor, Week 89 OLE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  Intracranial Tumor, Week 89 OLE |  |  |  |  | 1
  Lacunar Infarct, Week 89 OLE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  Lacunar Infarct, Week 89 OLE |  |  |  |  | 0
  Superficial Hemosiderosis, Week 89 OLE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  Superficial Hemosiderosis, Week 89 OLE |  |  |  |  | 0
  Territorial Infarct, Week 89 OLE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  Territorial Infarct, Week 89 OLE |  |  |  |  | 0
  Vasogenic Edema/Sulcal Effusion, Week 89 OLE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 360
  Vasogenic Edema/Sulcal Effusion, Week 89 OLE |  |  |  |  | 1

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 15 January 2021 (up to approximately 39 months)
Description: The safety-evaluable population included all participants who were randomly allocated and received at least one dose of study drug (semorinemab or placebo) during the double-blind treatment period with treatment groups defined according to actual treatment received.
Groups:
- Dose 2 Semorinemab Open Label: Semorinemab was administered intravenously at dose 2 in the open-label extension period.
Arm/Group | Placebo Double Blind Period | Dose 1 Semorinemab Double Blind Period | Dose 2 Semorinemab Double Blind Period | Dose 3 Semorinemab Double Blind Period | Dose 2 Semorinemab Open Label
All-Cause Mortality (participants affected / at risk) | 2/130 | 0/89 | 1/132 | 1/90 | 1/360
Serious Adverse Events (participants affected / at risk) | 14/130 | 17/89 | 17/132 | 16/90 | 17/360
Other Adverse Events (participants affected / at risk) | 76/130 | 57/89 | 88/132 | 60/90 | 76/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double Blind Period (N=130) | Dose 1 Semorinemab Double Blind Period (N=89) | Dose 2 Semorinemab Double Blind Period (N=132) | Dose 3 Semorinemab Double Blind Period (N=90) | Dose 2 Semorinemab Open Label (N=360)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double Blind Period (N=130) | Dose 1 Semorinemab Double Blind Period (N=89) | Dose 2 Semorinemab Double Blind Period (N=132) | Dose 3 Semorinemab Double Blind Period (N=90) | Dose 2 Semorinemab Open Label (N=360)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (7) | 10 (11) | 4 (4) | 5 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (9) | 8 (9) | 4 (5) | 3 (4)
Fatigue (General disorders) | 2 (2) | 1 (1) | 4 (5) | 5 (5) | 1 (3)
Nasopharyngitis (Infections and infestations) | 11 (15) | 5 (6) | 18 (24) | 12 (14) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 15 (21) | 6 (8) | 7 (8) | 5 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 10 (13) | 4 (4) | 10 (11) | 5 (8) | 10 (11)
Fall (Injury, poisoning and procedural complications) | 22 (26) | 14 (15) | 22 (33) | 7 (11) | 18 (21)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (6) | 10 (16) | 11 (15) | 6 (11) | 5 (5)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 5 (5)
Blood pressure increased (Investigations) | 2 (2) | 1 (1) | 8 (12) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 6 (7) | 10 (12) | 8 (8) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 8 (8) | 6 (7) | 5 (5)
Dizziness (Nervous system disorders) | 12 (12) | 5 (7) | 6 (7) | 7 (9) | 4 (4)
Headache (Nervous system disorders) | 10 (13) | 2 (2) | 8 (11) | 6 (9) | 15 (15)
Anxiety (Psychiatric disorders) | 3 (3) | 10 (10) | 6 (7) | 6 (6) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 5 (5) | 7 (8) | 5 (6) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 4 (4) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 7 (7) | 5 (8) | 5 (5)
Hypertension (Vascular disorders) | 7 (7) | 4 (4) | 14 (14) | 5 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT03289143/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03289143/SAP_001.pdf